CLINICAL TRIAL: NCT03274817
Title: A Proof of Concept Study of the Prevention of Mild Cognitive Impairment and Eventual Alzheimer's Disease Using F18 Flutemetamol
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-0228
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Depression; Escitalopram; Venlafaxine
MeSH Terms: conditions — Alzheimer Disease; Depression | interventions — Escitalopram; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Escitalopram (Active Comparator): Escitalopram (lexapro) is presently the most widely used selective serotonin reuptake inhibitor (SSRI) antidepressant.
  Interventions: Drug: Escitalopram Pill
- Venlafaxine (Active Comparator): Venlafaxine is a norepinephrine, serotonin and dopamine reuptake inhibitor antidepressant.The specific form of venlafaxine which will be employed is Effexor XR (venlafaxine hydrochloride extended release capsules)
  Interventions: Drug: Venlafaxine Pill
- Placebo (Placebo Comparator): Subjects randomized to group C will receive placebo tablets, which will be matched to the Lexapro and the Effexor XR as far as possible, and will also be administered on a once daily schedule at baseline.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Escitalopram Pill — Subjects randomized to group A will receive Lexapro (escitalopram), in an initial, baseline dosage of 5 mg daily.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Venlafaxine Pill — Subjects randomized to group B will receive Effexor XR (venlafaxine extended release capsules), in an initial baseline dosage of 37.5 mg daily.
  Other Names: Effexor XR
  Arms: Venlafaxine
Drug: Placebo Oral Tablet — Subjects randomized to group C will receive placebo tablets, which will be matched to the Lexapro and the Effexor XR as far as possible, and will also be administered on a once daily schedule at baseline.
  Arms: Placebo

SUMMARY:
This is an investigator-initiated study comparing two types of FDA-approved anti-depressants, Escitalopram and Venlafaxine, to placebo, in order to determine if these medications have positive effects on cognition and memory in those who are between the ages of 50 to 89 years old, who are cognitively normal, and who have subjective memory concerns. Research has shown that those who are cognitively normal but report subjective cognitive impairment are more likely to progress to mild cognitive impairment and Alzheimer's disease in the future. Anti-depressants such as Escitalopram and Venlafaxine have been shown to stimulate production of neurons in memory-sensitive areas such as the hippocampus. Therefore, the investigator is researching whether these drugs would help cognition in those with subjective cognitive impairment, and would help to prevent cognitive decline and eventual Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have subjective cognitive impairment (SCI) and be free of objective evidence of cognitive impairment. Operationally, this will be defined as subjects with Global Deterioration Scale (GDS) score of stage 2.4
* Subjects must be between 60 and 80 years of age.
* Subjects must have a knowledgeable informant (study partner) who can accompany them to the evaluations, or, when necessary, be available for telephone contact.
* Subjects must be otherwise healthy and fulfill all of the inclusion criteria for participation in the NYU ADC. Exclusion criteria are enumerated below.
* Subjects must be in a position to comply with all of the study procedures described herein.
* Subjects must have a minimum of 12 years of education.
* Subjects must be fluent in English.
* Subjects original language at birth and/or, in childhood, must have been English, alone, or in conjunction with other languages.

Exclusion Criteria:

* Subjects who have normal brain aging, who are free of subjective cognitive impairment (SCI), and are therefore categorized at GDS stage 1, will be excluded.
* Subjects with MCI or dementia and are therefore categorized as being at GDS stage 3 or greater, will be excluded.
* Subjects with a mini mental status examination (MMSE) score61 of ≤ 27 will be excluded.
* Subjects with a Hamilton Depression Scale (HDS) score ≥ 16,62 signifying the presence of notable depressive symptomatology which warrants treatment, will be excluded.
* Subjects with a primary diagnosis of depression or with a major depression diagnosis will be excluded.
* Subjects with a significant medical, neurologic, or psychiatric condition, including depression or anxiety disorder, that might interfere with cognition will be excluded.
* Subjects with a history of adverse reactions to escitalopram and/or venlaflaxine will be excluded.
* Subjects, who are judged to have had adverse reactions to selective serotonin reuptake inhibitor medications as a class, will be excluded.
* Subjects taking the antibiotic Zyvox (linezolid) or methylene blue therapy or who are planning to have a diagnostic procedure utilizing methylene blue dye, will be excluded.
* Subjects who are on psychoactive or cognitively active medications or who have received such medications in the prior 8 weeks, will be excluded. These excluded medications encompass antidepressant medications, antipsychotic medications, anxiolytic medications, cholinesterase inhibitors, memantine, antiseizure medications, antiparkinsonian medication and other CNS acting medications.
* Subjects who are receiving other medications or substances with reported neurogenic enhancer or neurogenic inhibitor effects will not be excluded. The reason for this inclusionary approach is that just as the effects of neurogenic enhancers on Alzheimer's disease appears to be complex (specifically, likely useful in prevention, possibly not useful effects on disease progression), the same complexity apparently applies to substances with reported neurogenic enhancer or inhibitor effects. For example, the angiotensin II receptor antagonist losartan has been reported to suppress running enhanced neurogenesis in the rat.63 This same medication and medication class has also been reported to be useful in improving memory64 and in the prevention of Alzheimer's disease, possibly by other mechanisms.65
* Subjects with a history of significant cerebrovascular disease will be excluded. This will be identified by one of the following:

  i. history of stroke. ii. Any focal signs of significant neuropathology from the neurological examination.

iii. A score of ≥ 4 on the Rosen modification of the Hachinski Ischemia Scale.66 iv. Focal pathology on the MRI scan, indicative of history of infarction. l. Past history of brain damage, seizure, mental retardation or serious neurological disorders.

* Significant history of alcoholism or drug abuse.
* Previous history of schizophrenia, mania, or major depression.
* Severe cardiac, pulmonary, vascular, metabolic, or hematologic conditions.
* Presence of a cardiac pacemaker.
* Presence of any metallic device or implant which would contraindicate an MRI (magnetic resonance imaging) scan of the brain.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Hostility or refusal to cooperate.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06-18 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Z-score for the hippocampal region of interest in the theta band | 24 Months
  responders show will less increase in score with treatment compared with baseline, in comparison with placebo treated subjects.
Multivariate Z score for overall theta abnormality in the frontal and parieto-temporal regions; | 24 Months
  Each subject can serve as their own control, z-transformed relative to initial values accessed for each of the endpoints. In addition, each subject can be evaluated relative to age-expected normal values.
Probability of deterioration from logistic regression predictive of future decline; | 24 Months
Z-score coherence (synchrony) between right central and parietal regions across all bands; | 24 Months
  Each subject can serve as their own control, z-transformed relative to initial values accessed for each of the endpoints. In addition, each subject can be evaluated relative to age-expected normal values.
Mean frequency across the total EEG brain spectrum. | 24 Months
Metabolic reduction in the hippocampal formation (a region including the hippocampal subiculum and the entorhinal cortex) assessed bilaterally. | 24 Months

SECONDARY OUTCOMES:
Brief Cognitive Rating Scale Axes I to V total scores | 24 Months
The Mini-Mental State Examination (MMSE) total scores | 24 Months
  30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia.
MAC-Q total score | 24 Months
  brief index of memory complaint.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Reisberg, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided